CLINICAL TRIAL: NCT03557645
Title: Hemodynamic Repercussions of Ventilator Hyperinflation Using Volume-controlled Ventilation: a Randomized Controlled Trial
Brief Title: Ventilator Hyperinflation and Hemodynamics
Acronym: VHI-HD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitário Augusto Motta (Other)
Collaborators: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: VHI Hemodynamics
Record Dates: First submitted 2018-05-13; First posted 2018-06-15 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Respiratory Failure; Respiratory Disorders
Keywords: mechanical ventilation; physiotherapy; ventilator hyperinflation; airway clearance technique
MeSH Terms: conditions — Respiratory Insufficiency; Respiration Disorders

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Baseline Mechanical Ventilation (Sham Comparator): The subjects will be kept in Volume Control Continuous Mandatory Ventilation (VC-CMV) with an inspiratory flow = 60Lpm and tidal volume = 6mL/IBW. Positive end-expiratory pressure and the inspired oxygen fraction will not be modified.
  Interventions: Device: Baseline Mechanical Ventilation
- VHI With Inspiratory Pause (Experimental): Application of a ventilator hyperinflation intervention with Volume Control Continuous Mandatory Ventilation (VC-CMV). The inspiratory flow will be set at 20Lpm, the tidal volume will be increased in steps of 200mL until the peak airway pressure of 40cmH2O is achieved, and an inspiratory pause will be applied at the end of inspiration. After achieving the target pressure, this ventilatory regimen will last 15 minutes. Positive end-expiratory pressure and the inspired oxygen fraction will not be modified.
  Interventions: Device: VHI With Inspiratory Pause
- VHI Without Inspiratory Pause (Experimental): Application of a ventilator hyperinflation intervention with Volume Control Continuous Mandatory Ventilation (VC-CMV). The inspiratory flow will be set at 20Lpm and the tidal volume will be increased in steps of 200mL until the peak airway pressure of 40cmH2O is achieved. After achieving the target pressure, this ventilatory regimen will last 15 minutes. Positive end-expiratory pressure and the inspired oxygen fraction will not be modified.
  Interventions: Device: VHI Without Inspiratory Pause

INTERVENTIONS:
Device: Baseline Mechanical Ventilation — The subjects will be kept in Volume Control Continuous Mandatory Ventilation (VC-CMV).
  Arms: Baseline Mechanical Ventilation
Device: VHI With Inspiratory Pause — Application of a ventilator hyperinflation intervention with Volume Control Continuous Mandatory Ventilation (VC-CMV) with an inspiratory pause.
  Arms: VHI With Inspiratory Pause
Device: VHI Without Inspiratory Pause — Application of a ventilator hyperinflation intervention with Volume Control Continuous Mandatory Ventilation (VC-CMV) without an inspiratory pause.
  Arms: VHI Without Inspiratory Pause

SUMMARY:
Ventilator hyperinflation (VHI) has been shown to be effective in improving respiratory mechanics, secretion removal, and gas exchange in mechanically ventilated patients; however, the literature is scarce concerning its safety and adverse effects. Thus, the aim of this study is to compare the hemodynamic repercussions of VHI in volume-controlled mode. In a randomized, controlled and crossover design, 24 mechanically ventilated patients will undergo 2 modes of ventilator hyperinflation (with and without an inspiratory pause) and a control intervention. Cardiac output, cardiac index, mean arterial pressure, pulmonary vascular resistance, systolic volume and other hemodynamic variables will be recorded during the interventions.

DETAILED DESCRIPTION:
Background: ventilator hyperinflation (VHI) has been shown to be effective in improving respiratory mechanics, secretion removal, and gas exchange in mechanically ventilated patients; however, the literature is scarce concerning its safety and adverse effects. Thus, the aim of this study is to compare the hemodynamic repercussions of VHI in volume-controlled mode.

Methods: in a randomized, controlled and crossover design, 24 mechanically ventilated patients will undergo 2 modes of ventilator hyperinflation (with and without an inspiratory pause of 2 seconds) and a control intervention. For the VHI interventions, the inspiratory flow will be set at 20 Lpm, and tidal volume will be increased until a peak pressure of 40cmH2O is achieved. During the control intervention, the patients will remain in volume-control ventilation with an inspiratory flow = 60Lpm and tidal volume = 6mL/IBW. The interval between interventions (washout) will be of 10 minutes or more, according to the time needed to recover the cardiac index to baseline values (maximum difference of 10%). Cardiac output, cardiac index, mean arterial pressure, pulmonary vascular resistance, systolic volume and other hemodynamic variables will be recorded during the interventions by using impedance cardiography.

ELIGIBILITY:
Inclusion Criteria:

* Patients under mechanical ventilation for more than 48h

Exclusion Criteria:

* mucus hypersecretion (defined as the need for suctioning < 2-h intervals),
* absence of respiratory drive,
* atelectasis,
* severe bronchospasm,
* positive end expiratory pressure > 10cmH2O,
* PaO2-FiO2 relationship < 150,
* mean arterial pressure < 60mmHg,
* inotrope requirement equivalent to >15 ml/h total of adrenaline and noradrenalin,
* intracranial pressure > 20mmHg

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-11-05 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Cardiac Output | Baseline (before) and 10 minutes after the onset of VHI modesBasel
  Estimation of cardiac output variation using thoracic bioimpedance

SECONDARY OUTCOMES:
Change in Cardiac Index | Baseline (before) and 10 minutes after the onset of VHI modes
  Estimation of cardiac index variation using thoracic bioimpedance
Change in Vascular pulmonary resistance | Baseline (before) and 10 minutes after the onset of VHI modes
  Estimation of vascular pulmonary resistance variation using thoracic bioimpedance
Change in Systolic Volume | Baseline (before) and 10 minutes after the onset of VHI modes
  Estimation of systolic volume variation using thoracic bioimpedance
Change in Mean Arterial Pressure | Baseline (before) and 10 minutes after the onset of VHI modes
  Recording of mean arterial pressure variation using an automatic noninvasive device
Change in Cardiac Output II | Baseline (before) and 5 minutes after the end of VHI modes
  Estimation of cardiac output variation using thoracic bioimpedance
Change in Cardiac Index II | Baseline (before) and 5 minutes after the end of VHI modes
  Estimation of cardiac index variation using thoracic bioimpedance
Change in Vascular pulmonary resistance II | Baseline (before) and 5 minutes after the end of VHI modes
  Estimation of vascular pulmonary resistance variation using thoracic bioimpedance
Change in Systolic Volume II | Baseline (before) and 5 minutes after the end of VHI modes
  Estimation of systolic volume variation using thoracic bioimpedance
Change in Mean Arterial Pressure II | Baseline (before) and 5 minutes after the end of VHI modes
  Recording of mean arterial pressure variation using an automatic noninvasive device

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Guimaraes, PhD, Study Chair — Centro Universitário Augusto Motta
Locations (1):
- Hospital Santa Martha, Niterói, Rio de Janeiro, Brazil

REFERENCES:
- [Result] Berney S, Denehy L. A comparison of the effects of manual and ventilator hyperinflation on static lung compliance and sputum production in intubated and ventilated intensive care patients. Physiother Res Int. 2002;7(2):100-8. doi: 10.1002/pri.246. PMID 12109234
- [Result] Lemes DA, Zin WA, Guimaraes FS. Hyperinflation using pressure support ventilation improves secretion clearance and respiratory mechanics in ventilated patients with pulmonary infection: a randomised crossover trial. Aust J Physiother. 2009;55(4):249-54. doi: 10.1016/s0004-9514(09)70004-2. PMID 19929767
- [Result] Anderson A, Alexanders J, Sinani C, Hayes S, Fogarty M. Effects of ventilator vs manual hyperinflation in adults receiving mechanical ventilation: a systematic review of randomised clinical trials. Physiotherapy. 2015 Jun;101(2):103-10. doi: 10.1016/j.physio.2014.07.006. Epub 2014 Oct 6. PMID 25453540
- See also: Main researcher - personal profile in Researchgate — https://www.researchgate.net/profile/FERNANDO_GUIMARAES